CLINICAL TRIAL: NCT04769791
Title: Three Inflation Methods of the Laryngeal Mask Airway Ambú Auraonce™ and Its Pharyngolaryngeal Adverse Effects
Brief Title: Three Inflation Methods of the Ambú Auraonce™ and Its Adverse Effects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Principal Investigator, Teresa Prim, Principal investigator, Instituto de Investigación Hospital Universitario La Paz
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Idipaz 4888
Record Dates: First submitted 2021-02-12; First posted 2021-02-25 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Laryngeal Mask Airway
Keywords: laryngeal mask; intracuff pressure; sore throat
MeSH Terms: conditions — Pharyngitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- cuff inflation by the residual volume (Experimental): LMA will be inserted with the initial inflating volume correspondent to residual volume group ( RV group): volume result of equilibrating pressure between intracuff pressure and atmospheric pressure. A 20 ml syringe without plunger is connected to the laryngeal cuff for 5 minutes.
  Interventions: Device: intracuff pressure measurement
- cuff inflation by half of the maximum volume (Experimental): LMA will be inserted with the initial inflating volume correspondent to half of the maximum volume recommended by manufacturers (MV group):
  Interventions: Device: intracuff pressure measurement
- unchanged cuff inflation volume (Experimental): LMA will be inserted with the initial inflating volume correspondent to unchanged volume group (NV group): LMA is unpacked and used without inflating or deflating the cuff.
  Interventions: Device: intracuff pressure measurement

INTERVENTIONS:
Device: intracuff pressure measurement — intracuff pressure is measured by a pressure manometer
  Arms: cuff inflation by the residual volume
Device: intracuff pressure measurement — intracuff pressure is measured by a pressure manometer
  Arms: cuff inflation by half of the maximum volume
Device: intracuff pressure measurement — intracuff pressure is measured by a pressure manometer
  Arms: unchanged cuff inflation volume

SUMMARY:
Laryngeal mask airway device (LMA) is a common device used in the daily practice for airway management. Consecutive generations have permitted an expansion of its use, probably because of a rapid increase of ambulatory surgical procedures and also due to the development of procedures in areas away from the operating room.

The cuff inflating volume is not standardized and it is common practice to inflate the LMA cuff according to the manufacturer's recommendations, without using a manometer.

A hyperinflation of the LMA cuff was associated with complications ranging from sore throat, or dysphagia and dysphonia, to more serious complications such as paralysis of the vocal cord, arytenoid cartilages dislocation, recurrent laryngeal nerve injury and hypoglossal nerve injury. Also, the excess of volume or pressure is related to poor ventilation and increase the risk of gastric insufflation.

The aim of this study is to evaluate the best cuff inflation method, in order to limit the intracuff pressure beyond the recommended maximum pressure (PM < 60 cmH2O) and to allows decrease the pharyngo-laryngeal complications.

The Primary outcome is to compare three different cuff inflating methods using AuraOnce™ LMA during fibrobronchoscopy and endobronchial ultrasound (EBUS) procedures, and to control the intracuff pressure, and the effect on pharyngo-laryngeal complications.

The three different cuff inflating methods are: 1) residual volume group (RV group) 2) half of the maximum volume group (MV group) 3) unchanged volume group (NVgroup)

DETAILED DESCRIPTION:
This is a prospective randomized controlled trial. The study was approved by the Ethics Committee of University Hospital of La Paz, Madrid. Written informed consent will be obtained from each patient before the procedure. We plan to include 210 patients scheduled for a fibrobronchoscopy with EBUS-transbronchial needle aspiration (TBNA) procedures under general anesthesia using a LMA. Patients will be allocated randomly to one of three groups of cuff inflating methods according to computer-generated randomization. The size of LMA will be chosen according to body weight, following the manufacturer recommendations (LMA size 3 for patients of 30-50 kg, LMA size 4 for patients of 50-70 kg and LMA size 5 for patients with a weight >70 kg). After standard monitoring with electrocardiography, noninvasive blood pressure device and pulse oximeter were applied, general anesthesia will be induced with Propofol 2.5 mg.kg-1 and fentanyl 1 mcg.kg-1 intravenously Face mask ventilation with 100% oxygen will be used after patients have lost eyelash reflex. Then, the assigned LMA will be inserted, after appropriate conditions for insertion are obtained. LMA Insertion will be performed with standard maneuver according to LMA practice manual by the same experienced anesthesiologist (> 1-year use experience). The initial position of LMA will be assessed by visualization of bilateral chest movement when positive pressure ventilation will be performed and the square capnography waveform is observed on the monitor screen.

If the LMA is not in the proper position at the first attempt, we will use an "up and down" maneuver to adjust and reposition LMA to attain satisfactory ventilation. If this maneuver fails, LMA will be withdrawn from the mouth of the patients and a second attempt will be authorized to acquire a correct position. If the proper position of LMA cannot be achieved after two attempts, the airway will be controlled with another device or a tracheal intubation will be performed and the patients will be excluded from the trial.

The patient´s lungs will be ventilated with the anesthesia machine in controlled volume mode, using the following parameters: Tidal volume, 8 ml/kg; frequency, 12-14 per min; the ratio of inspiratory and expiratory, (I: E) = 1:2; and positive end expiratory pressure, 5 cmH20.

After the LMA will be fixed with adhesive tape and the vital signs will be stable, the LMA cuff will be connected with a closed system manometer composed of a three-way stopcock, a 5 ml syringe and a manometer. Intracuff pressure will be measured and recorded, if it exceeds of 60 cmH20 we will deflate the cuff 1 mL by 1 mL with the syringe until intracuff pressure reaches 60 cmH20. The deflated volume and the final intracuff pressure will be recorded. We will measure the inspiratory peak airway pressure, the volume difference of inspiratory and expiratory tidal volume under the positive pressure ventilation. The plateau pressure, medium pressure and Compliance will also be recorded at the corresponding cuff inflating volume, before and after measuring OLP. The OLP will be measured simultaneously at the corresponding cuff inflating volume, by setting the airway pressure relief valve (APL) of the breathing circuit to 40 cmH20 at a fixed gas flow rate of 4 L/ min and reading the airway pressure on manometer at which equilibrium of airway pressure will be established or at the pressure the air leakage will be heard.

Fiberoptic visibility scores will be recorded on a scale of 1 to 4 (4: only vocal cords visible, 3: vocal cords plus posterior epiglottis visible, 2: vocal cords plus anterior epiglottis visible, 1: vocal cords not seen). A score of 1 will be considered the worst and a score of 4 was considered the best.

Any adverse events (i.e., desaturation (pulse oximetry< 90%), aspiration/regurgitation, bronchospasm, airway obstruction, coughing, gagging or vomiting) and corresponding interventions will be recorded.

After the procedure, all patients will be transferred to the recovery unit and observed for at least 1 hour. Observed adverse effects, such as sore throat, hoarseness, aphasia, nausea and vomiting will be recorded in the recovery room period.

At 24h, a home telephone interview will record these parameters, as well as patient satisfaction scores using visual analog scales.

ELIGIBILITY:
Inclusion Criteria:

* Patients age between 18 and 90 years
* American Society of Anesthesiologists (ASA) physical status I-III
* fiberoptic bronchoscopy procedure and EBUS-TBNA procedure programmed.
* Fasted for 6 hours before procedure.
* Management of the airway for the same anesthetic.
* Use de laryngeal mask airway for boarding and maintenance of airway permeability

Exclusion Criteria:

* LMA is contraindicated because high risk of aspiration (full stomach, gastroesophageal reflux history, pregnant)
* predictors of difficult airway such restricted mouth opening (< 3 cm of interincisal distance)
* patients with any pathology of the neck, upper respiratory or upper alimentary tract
* BMI > 40 Kilogram / m2
* dysphagia o hoarseness

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2018-11-21 (Actual); Study Completion 2018-11-21 (Actual)

PRIMARY OUTCOMES:
Intracuff Pressure | procedure ( after correct placement of SGD)
  Compare Intracuff Pressure of three different cuff inflating volume methods with laryngeal mask, to control the intracuff pressure

SECONDARY OUTCOMES:
time of insertion | procedure ( from pick up to correct placement of SGD
  Compare time of insertion in the three different cuff inflating volume methods
insertion attempts | procedure ( from pick up to correct placement of SGD
  Compare insertion attempts in the three different cuff inflating volume methods
OLP | procedure ( after correct placement of SGD)
  We measure the oropharyngeal leak pressure (OLP) as a sealing efficacy test.
positioning of the LMA | procedure (after correct placement of SGD)
  Compare the positioning of the LMA with the three methods of inflating cuff. Fiberoptic visibility scores will be recorded on a scale of 1 to 4 (4: only vocal cords visible, 3: vocal cords plus posterior epiglottis visible, 2: vocal cords plus anterior epiglottis visible, 1: vocal cords not seen). A score of 1 will be considered the worst and a score of 4 was considered the best.
pharyngolaryngeal complications | day 2
  Describe sore throat, dysphagia and dysphonia

CONTACTS AND LOCATIONS:
Overall Officials: TERESA PRIM MARTINEZ, MD, Principal Investigator — HOSPITAL La Paz
Locations (1):
- Teresa Prim Martinez, Madrid, Spain

REFERENCES:
- [Background] Seet E, Yousaf F, Gupta S, Subramanyam R, Wong DT, Chung F. Use of manometry for laryngeal mask airway reduces postoperative pharyngolaryngeal adverse events: a prospective, randomized trial. Anesthesiology. 2010 Mar;112(3):652-7. doi: 10.1097/ALN.0b013e3181cf4346. PMID 20179502
- [Background] Ghai B, Sethi S, Ram J, Wig J. Cuff filling volumes for pediatric classic laryngeal mask airways: comparison of clinical end points versus adjusted cuff pressure. Paediatr Anaesth. 2013 Feb;23(2):122-6. doi: 10.1111/pan.12023. Epub 2012 Sep 18. PMID 22985184
- [Background] Keller C, Puhringer F, Brimacombe JR. Influence of cuff volume on oropharyngeal leak pressure and fibreoptic position with the laryngeal mask airway. Br J Anaesth. 1998 Aug;81(2):186-7. doi: 10.1093/bja/81.2.186. PMID 9813520
- [Background] Li BB, Yan J, Zhou HG, Hao J, Liu AJ, Ma ZL. Application of Minimum Effective Cuff Inflating Volume for Laryngeal Mask Airway and its Impact on Postoperative Pharyngeal Complications. Chin Med J (Engl). 2015 Oct 5;128(19):2570-6. doi: 10.4103/0366-6999.166034. PMID 26415792
- [Background] Ruananukun N, Watcharotayangul J, Jeeranukosol S, Komonhirun R. Correlation and variation of cuff inflating volumes and pressures in different adult models of laryngeal mask: a prospective randomized trial. BMC Anesthesiol. 2020 May 7;20(1):108. doi: 10.1186/s12871-020-01028-4. PMID 32380954
- [Derived] Prim T, Brogly N, Guasch E, Diez J, Gilsanz F. Efficacy and safety of three inflation methods of the laryngeal mask airway Ambu(R) Auraonce: a randomized controlled study. J Clin Monit Comput. 2024 Feb;38(1):37-45. doi: 10.1007/s10877-023-01061-x. Epub 2023 Aug 4. PMID 37540323